CLINICAL TRIAL: NCT02336672
Title: EUS-Guided Cryothermal Ablation in Patients With Stage III (Locally Advanced and Borderline Resectable) Pancreatic Adenocarcinoma
Brief Title: EUS-Guided Cryothermal Ablation in Patients With Stage III Pancreatic Adenocarcinoma (HybridTherm Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Paolo Giorgio Arcidiacono, MD, Head of Pancreatico-Biliary and Endosonography Division, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTP/2014
Record Dates: First submitted 2014-12-16; First posted 2015-01-13 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Adenocarcinoma Non-resectable
Keywords: Pancreatic adenocarcinoma; Cryothermoablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A Chemotherapy (No Intervention): Patients receiving chemotherapy alone. These patients start standard chemotherapy right after the oncologist's evaluation according to accepted Guidelines of the Italian Association of Medical Oncologists (AIOM). Restaging is performed 2, 4 and 6 months after chemotherapy onset, with MDCT scan and DW-MRI.
- Group B Chemotherapy + HybridTherm (Experimental): Patients receiving chemotherapy plus EUS-guided Cryothermal Ablation with HybridTherm probe. These patients are first treated by cryothermal ablation and one week after they start with chemotherapy. Cryothermal ablation can be performed up to three times, with interval of 4 +/- 1 weeks. Restaging is performed 2, 4 and 6 months after chemotherapy onset, with MDCT scan and DW-MRI.
  Interventions: Device: Cryothermal ablation

INTERVENTIONS:
Device: Cryothermal ablation — Procedures are performed with patients sedated by anaesthesiologists. Device setting and application time are set and recorded on a computer, that analyzes the changes of the tissue's properties. The setting of the maximal application time is based on the results of our previously described ex-vivo and in-vivo studies and is adjusted to the tumour's size, thus ensuring a reduction of procedure-related complications. Application of Power Doppler makes the procedure safer. The HybridTherm probe is guided under real-time EUS into the tumour, and the success of its placement is an index of the treatment's feasibility. The system analyzes the effects on the tissue and EUS records the changes of the tissue, the growing edema around the treated area, and the tissue devitalization.
  Other Names: HybridTherm probe
  Arms: Group B Chemotherapy + HybridTherm

SUMMARY:
In patients with locally advanced tumour, neoadjuvant treatment has been proposed in various modalities as a way to decrease size and downstage the tumour leading to a re-sectable disease. The HybridTherm probe (HTP), (ERBE Elektromedizin GmbH, Tübingen, Germany) combines bipolar RF-ablation with cryogenic induced cooling. A bipolar radiofrequency system creates ablation with less collateral thermal damage than standard monopolar systems but with the trade-off to lose overall efficiency.

DETAILED DESCRIPTION:
About 40% of patients with pancreatic cancer have no metastasis at the moment of diagnosis, but in 20% of patients surgery is not feasible due to vascular invasion or poor general conditions. These patients with stage III pancreatic cancer (locally advanced or borderline resectable) may benefit from neoadjuvant chemotherapy or chemoradiotherapy. The HybridTherm probe is a new, minimally invasive device that can be safely applied under EUS guidance to locally ablate the pancreatic tissue adding a local efficacy to the systemic activity offered by chemotherapy and could give these patients a bigger chance of survival. The present study is an interventional randomized controlled phase II/III trial (device), that assigns patients into two groups: patients receiving standard chemotherapy alone and those receiving chemotherapy plus EUS-guided HybridTherm ablation. The randomization is performed at the time of EUS diagnosis and staging.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnosis
* patients with borderline resectable/locally advanced pancreatic adenocarcinoma;
* patients no previously treated with neoadjuvant treatments, irrespective of the regimen
* age >18 years; ≤ 80
* genders eligible for study: both
* patients who can express their consent
* Karnofsky Performance status >70;
* Life expectancy >6 months.
* PLT>100000/mcl; INR<1.5.
* adequate renal function with a creatinine threshold
* adequate bone marrow function (WBC ≥3500)

Exclusion Criteria:

* pregnancy
* acute pancreatitis
* patients having distant metastasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 6-months after therapy onset
  To demonstrate the efficacy of the HybridTherm probe in the control of the tumour progression in terms of progression-free survival, measured at 6-month after ther-apy onset (PFS-6). PFS-6 takes in consideration the tumor growth in relation to the volume/size evaluated as a difference between the previous and the current examination. In practice, it is the time interval between the enrolment of the patient and the first radiological evidence of tumor progression.
  For patients who were resected (R0 and R1) the PFS is the time until the first radio-logical evidence of tumor recurrence, regardless size.
  For not resected patients the PFS is the time until the first radiological evidence of a growth of the lesion > 20% in comparison to the previous exam.

SECONDARY OUTCOMES:
Response to treatment | At 2 and 4 months after the treatment
  Evaluated by the radiological response to the treatment calculated on the differ-ences of radiological images (DW-MRI) before treatment onset and after two and four month of treatment
Evaluation of cell disruption / necrosis of the treated area | At 2 and 4 months after the treatment
  Measured with the Apparent Diffusion Coefficient in the dw-MRI which will be per-formed at the time of patients' enrolment, after HTP treatment (Group B) and after two and four month of treatment.
Rate of resectability | After 4 months pf treatment
  Evaluated by the number of resectable patients after four month of treatment
R0 Resection Rate: | After surgical resection
  Evaluated by the number of R0 resections for those patients who were submitted to sur-gery (see Rate of resectability) on the basis of the pathologists finding

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Giorgio Arcidiacono, MF FASGE, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Ospedale San Raffaele Irccs, Milan, MI, Italy